CLINICAL TRIAL: NCT01247948
Title: A Multi-center Randomized Controlled Trial Evaluating the Accuracy of Navigation Assisted Pedicle Screw Placement of Spine Surgery
Brief Title: Evaluating the Accuracy of Navigation Assisted Pedicle Screw Placement of Spine Surgery
Acronym: J0001I41
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Tian Wei ,director of the hospital, Beijing Jishuitan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: jst2010caos; jstssrct001 (Other: Beijing Jishuitan Hospital)
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-11

CONDITIONS: Pedicle Screw of Fixation
Keywords: pedicle screw of fixation operation; spine surgery; navigation assisted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- navigation assisted spine surgery (Experimental)
  Interventions: Procedure: navigation assisted spine surgery; Procedure: traditional spine surgery

INTERVENTIONS:
Procedure: navigation assisted spine surgery — navigation assisted pedicle screw placement of spine surgery
  Other Names: navigation assisted pedicle screw placement of spine surgery
Procedure: traditional spine surgery — traditional spine surgery without navigation assist
  Other Names: traditional spine surgery without navigation assist

SUMMARY:
The purpose of this study is to investigate the difference of the accuracy and safety between traditional spine surgery and computer assisted navigation system spine surgery.

DETAILED DESCRIPTION:
The object of study is the patients who are going to undergo pedicle screw fixation operation. there are two clinical trial centers.one is beijing jishuitan hospital,the other is beijing shuili hospital.the study protocol will be reviewed by the Ethics Committee of Beijing Jishuitan Hospital. after the patients sign the informed consent,they will be divided into two groups randomly.the patients' basic information and medical informations including the accuracy and safety will be collected.the data above all will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients who need to undergo pedicle screw fixation surgery
* Sign informed consent
* Capacity person

Exclusion Criteria:

* refused to sign the informed consent
* the age is not between 18 and 75 years old

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-12 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
the accuracy of pedicle screw | one week after the spine surgery
  one week after the spine surgery,measure the accuracy of pedicle screw by CT examination

SECONDARY OUTCOMES:
complication | three days after the spine surgery
  the complication would be recorded three days after the spine surgery

CONTACTS AND LOCATIONS:
Overall Officials: Wei Tian, doctor, Study Chair — Beijing Jishuitan Hospital